CLINICAL TRIAL: NCT06983080
Title: The Efficacy of Trazodone for the Treatment of Insomnia in Older Adults: A Randomized Controlled Trial (The TRADITION Study)
Brief Title: Efficacy of Trazodone to Treat Insomnia in Older Adults (TRADITION Study)
Acronym: TRADITION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-12893
Record Dates: First submitted 2025-03-27; First posted 2025-05-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Insomnia Chronic; Older People; Drug Therapy
Keywords: insomia; Trazodone; Older adults; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crossover Trazodone then Placebo arm (Experimental): Participants will receive 25 to 50 mg of trazodone once daily at bedtime for 28 days. After a 14-day washout period, participants will receive a placebo for another 28 days.
  Interventions: Drug: Trazodone 25 mg
- Crossover Placebo then Trazodone arm (Experimental): Participants will receive a placebo once daily at bedtime for 28 days. After a 14-day washout period, participants will receive 25 to 50 mg of trazodone for another 28 days.
  Interventions: Drug: Trazodone 25 mg

INTERVENTIONS:
Drug: Trazodone 25 mg — Trazodone 25 mg at bedtime, which can be increased to 50 mg after 14 days of treatment.

SUMMARY:
This study aims to evaluate how effective trazodone is in treating insomnia in adults aged 65 years and older. The main question it aims to answer is :

- Is trazodone more effective than a placebo in reducing the severity of insomnia symptoms in older adults?

Participants will :

* Take 25 to 50 mg of trazodone or a matching placebo before bed for 28 days. After a 2-week break, they will then take the other medication for another 28 days.
* Visit the clinic three times for checkup and test
* Complete a sleep diary and wear an actimeter during the night.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 or older in an outpatient setting
* Insomnia according to the criteria of the ICSD-3R

Exclusion Criteria:

* Contraindication to trazodone (hypersensitivity)
* Presence of a ventricular cardiac arrhythmia (e.g., torsades de pointes)
* Recent myocardial infarction (< 6 months)
* Substances that may alter sleep (hypnotics or any other medication intended to induce sleep, such as mirtazapine or quetiapine, corticosteroids, melatonin, psychostimulant drugs)
* Active, unstable psychiatric disorder
* Initiation or titration of an antidepressant within the past 6 months
* Cognitive-behavioral therapy ongoing or planned during the study period
* Major neurocognitive disorder (NCD) moderate or severe, or other cognitive disorders that may prevent the participant from being able to participate in the study, according to the judgment of the evaluating physician
* Parkinson's disease
* Priapism
* Known angle-closure glaucoma
* Symptomatic restless leg syndrome > 3 times per week
* QTc interval > 500 ms
* Parasomnias, dyssomnias other than insomnia
* Severe sleep apnea with AHI > 30 without CPAP treatment
* Use of a monoamine oxidase inhibitor
* Use of a strong CYP 3A4 inducer or inhibitor
* Hospitalized individuals
* Seizure within the past 6 months
* History of orthostatic hypotension
* History of delirium within the last 6 months
* Consumption of > 14 alcoholic drinks per day or use of alcohol to induce sleep.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | At baseline or at day 1, at day 36 and at day 77.
  The ISI is a self-assessment questionnaire that evaluates the nature, severity, and impact of insomnia. The typical recall period is the past month. The dimensions assessed are: the severity of falling asleep, maintaining sleep, and waking up too early in the morning; sleep dissatisfaction; the interference of sleep difficulties with daytime functioning; the visibility of sleep problems to others; and the distress caused by sleep difficulties. A 5-point Likert scale is used to evaluate each item. The total score is interpreted as follows: no insomnia 0-7; subclinical insomnia 8-14; moderate insomnia 15-21; and severe insomnia 22-28. It is increasingly used as a measure of treatment response in clinical research. Data confirm its reliability and the validity of the measurements obtained in the older adult population.

SECONDARY OUTCOMES:
Insomnia daytime symptoms and Impacts Questionnaire | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The IDSIQ is a questionnaire covering 14 different items that specifically measures the impact of insomnia on various aspects of daytime functioning. The questions are grouped into three areas, each representing the main daytime symptoms and impacts of insomnia on drowsiness (four items), alertness/cognition (six items), and mood (four items). Each item is rated on an 11-point numerical scale (from 0 to 10), with lower scores indicating better daytime functioning. It has been found to be sensitive to changes in patients experiencing daytime effects. It is quick to administer, easy to complete, and has reliable reproducibility (test-retest). It can be used in clinical trials to assess changes and the effectiveness of a treatment on daytime functioning and for the recording of new drugs for insomnia. Regulatory authorities now require that the effectiveness of clinical trials for medical products against insomnia be measured not only by treating physicians but also by the p
Subjective Sleep onset latency | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  Subjective time duration, in minutes, between the time the participant attempts to fall asleep (e.g., lights off, lying in bed) and the time they perceive they have fallen asleep.
Subjective wake after sleep onset | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The perceived total duration, in minutes, of all periods of wakefulness occurring after initial sleep onset and before final awakening
Subjective Total sleep time | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The perceived total duration, in minutes, of actual sleep obtained during the night, excluding periods of wakefulness.
Subjective sleep efficiency | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The perceived percentage of time spent asleep while in bed, calculated as the ratio of subjective total sleep time (sTST) to time in bed (TIB), multiplied by 100
Objective sleep onset latency | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The estimated duration, in minutes, between the time the participant attempts to fall asleep (e.g., lights out or bedtime) and the onset of the first sustained period of sleep, as detected by actigraphy
Objective Wake After Sleep Onset | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The estimated total duration, in minutes, of wakefulness occurring after the initial sleep onset and before final awakening, as detected by actigraphy
Objective Total Sleep Time | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The estimated total duration, in minutes, of actual sleep obtained during the sleep period, as detected by actigraphy, excluding all periods of wakefulness
Objective Sleep Efficiency | At baseline daily from day 1 to day 7, and during 7 days the first and last week of each treatment
  The estimated percentage of time spent asleep while in bed, calculated as the ratio of objective total sleep time (oTST) to objective time in bed (oTIB), multiplied by 100 as measured by actigraphy.
Adverse events | At Day 36 and day 77
  Incidence of at least one adverse event. Incidence of severe adverse events. Proportion of participants who discontinued due to adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is no need since it is a single center study.